CLINICAL TRIAL: NCT06008249
Title: A Multi-arm, Adaptive, Group-sequential Trial NETwork to Evaluate Drug Efficacy in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Platform Trial to Assess the Efficacy of Multiple Drugs in Amyotrophic Lateral Sclerosis (ALS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting TRICALS Foundation (Other)
Collaborators: Fight MND (Unknown); Research Foundation Flanders (Other); MNDA (Unknown); Thierry Latran Foundation (Unknown); Ulla-Carin Lindquist Foundation (Unknown); Luzon Foundation (Unknown); Alan Davidson Foundation (Unknown); My name'5 Doddie Foundation (Unknown); Stichting ALS Nederland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAGNET
Record Dates: First submitted 2023-08-14; First posted 2023-08-23 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Lithium Carbonate

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 2:1 ratio to receive either lithium carbonate or placebo
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium carbonate (Experimental): Lithium carbonate 400 mg capsules will be taken once daily, starting with one capsule (400 mg daily) initially titrated up to two or three capsules daily, depending on blood lithium levels. The target range for the lithium plasma level will be between ≥0.4 mmol/l and ≤ 0.8 mmol/l. Maximum duration is 24 months.
  Interventions: Drug: Lithium Carbonate 400 MG
- Placebo (Placebo Comparator): Patients start with 1 capsule to be taken once daily, with subsequent sham dose adjustments made to patients on placebo to maintain blinding in clinical sites.
  Interventions: Drug: Lithium Carbonate 400 MG

INTERVENTIONS:
Drug: Lithium Carbonate 400 MG — Lithium carbonate vs placebo (2:1)

SUMMARY:
The objective of this phase III, placebo-controlled platform study is to investigate the efficacy of drugs for patients with ALS (Amyotrophic lateral sclerosis).

DETAILED DESCRIPTION:
This study uses an innovative multi-arm, adaptive trial design to investigate the efficacy of multiple treatments simultaneously. Currently one study-arm is active, investigating the efficacy and safety of lithium carbonate versus placebo in patients with ALS. Only patients with a specific UNC13A genotype (approximately 1 in 6 ALS patients) are eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years at the time of screening.
2. Diagnosis of ALS according to the revised El Escorial criteria (possible, probable-laboratory supported, probable or definite).
3. Capable of providing informed consent and complying with trial procedures, including randomization to sub-studies.
4. TRICALS risk profile > -6.0 and < -2.0 **
5. The use of riluzole will be permitted during the study. Subjects taking riluzole must be on a stable dose for at least 30 days prior to the baseline visit, or stopped taking riluzole at least 30 days prior to the baseline visit.
6. Women of childbearing potential* must have a negative pregnancy test at baseline and be non-lactating.
7. Men must agree to practice contraception for the duration of the trial and for at least 3 months after last dose of study drug.
8. Men must not plan to father a child or to provide sperm for donation for the duration of the trial and 3 months after the last dose of study drug.
9. Women must not be able to become pregnant (e.g. post-menopausal***, surgically sterile or using effective birth control methods) for the duration of the study. Effective contraceptives are defined as having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label, including: abstinence, hormonal contraception, intrauterine device in place for ≥ 3 months Appendix 1). Women of childbearing potential must have a negative pregnancy test at baseline, and be non-lactating. Women who are pregnant or are actively seeking to become pregnant, and women of reproductive potential who are not using effective contraceptives are excluded.

Exclusion Criteria:

1. Laboratory Criteria at baseline:

   * ALT (alanine transaminase) ≥ 5 times upper limit of normal (ULN)
   * AST (aspartate aminotransferase) ≥ 3 times ULN
   * Bilirubin ≥ 1.5 times ULN
   * Estimated glomerular filtration rate (eGFR) < 50 mL / min / 1.73 m2 based on Cystatin C, if not available eGFR can also be calculated based on creatinine clearance.
   * Platelet concentration of < 100 x109 per L
   * Absolute neutrophil count of < 1x109 per L
   * Haemoglobin < 100 g/L (<6.2 mmol/L)
   * Amylase & lipase ≥ 2 times ULN (suspected pancreatitis)
   * Lactate ≥ 2 times ULN (suspected lactate acidosis)
2. Moderate to severe hepatic impairment according to Child-Pugh classification (Class B or higher; score ≥ 7). Child-Pugh classification is based on bilirubin, albumin, International Normalized Ratio (INR) and presence of encephalopathy or ascites.
3. Participation in any other investigational drug trial or using investigational drug (within 30 days prior to screening).
4. Hypothyroidism unresponsive to thyroid hormone supplementation.
5. Subjects using non-invasive ventilation (NIV, ≥22 h per day) or having a tracheostomy.
6. Subjects taking edaravone within 30 days prior to screening. Edaravone is approved by the FDA, but remains an investigational product in Europe and Australia.
7. Clinically significant history of unstable or severe cardiac (e.g. congestive heart failure, coronary insufficiency and arrhythmias), oncological, hepatic or renal disease, neuromuscular diseases, significant pulmonary disorder or other medically significant illness.
8. Drug or alcohol abuse.
9. Unstable psychiatric illness defined as psychosis or untreated major depression within 90 days of the screening visit. This exclusion criterion is based on a prior psychiatric diagnosis that is unstable as determined by the subject's treating Psychiatrist.
10. Presence of frontotemporal dementia which prevents informed consent.

Lithium carbonate study-specific exclusion criteria:

1. Patients heterozygous or homozygous for the A-allele of rs12608932 (UNC13A)
2. Known allergy or hypersensitivity to lithium, or its excipients, or to the components of the placebo.
3. Brain injury with posttraumatic epilepsy or neurologic deficit, excluding a concussion in the medical history. Brain infarction is an exclusion criterion, a transient ischemic attack is not.
4. Addison disease.
5. Patients with the following co-medication: antipsychotics, digoxin and calcium antagonists, carbamazepine, methyldopa, verapamil and diltiazem.
6. Brugada Syndrome or family history of Brugada Syndrome.
7. Plasma sodium <120 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival, defined as time to death from any cause or respiratory insufficiency (DRI; defined as tracheostomy or the use of non-invasive ventilation for ≥22 h per day for ≥10 consecutive days) | endpoint or 24 months
  A tracheostomy for ventilation is meant here

SECONDARY OUTCOMES:
Composite endpoint evaluating daily functioning and survival based on the joint model framework of survival and longitudinal ALSFRS-R total scores | endpoint or 24 months
  The ALSFRS-R (Amyotrophic Lateral Sclerosis Rating Scale-revised) is a 12 item participant self-report measure that monitors ALS disease progression, where a higher score reflects a better outcome.
Daily functioning, defined as mean change from baseline in ALSFRS-R total score. | endpoint or 24 months
  The ALSFRS-R (Amyotrophic Lateral Sclerosis Rating Scale-revised) is a 12 item participant self-report measure that monitors ALS disease progression, where a higher score reflects a better outcome.
Respiratory function, defined as mean change from baseline in SVC (%predicted of normal according to the GLI-2012 reference standard) | endpoint or 24 months
  Slow vital capacity (SVC) is measured in litres, and as a % of predicted. A higher score reflects a better outcome.
Quality of life, defined as change from baseline on the EQ-5D Visual Analogue Scale (single-item scale) | endpoint or 24 months
  The EQ-5D-5L (EuroQol 5 Dimension 5 Level) questionnaire is a standardised measure of health-related Quality of Life, using a Visual Analogue Scale. A higher score relates to a better outcome
Quality of life, defined as change from baseline on the EQ-5D | endpoint or 24 months
  The EQ-5D-5L (EuroQol 5 Dimension 5 Level) questionnaire is a standardised measure of health-related Quality of Life. A lower score relates to a better outcome
Neuropsychological status, defined as change from baseline on the ECAS | endpoint or 24 months
  ECAS (Edinburgh Cognitive and Behavioral Amyotrophic Lateral Sclerosis Screen) is a multidomain assessment questionnaire used in ALS to assess cognitive and behavioural changes where a higher score relates to a better outcome.
Neuropsychological status, defined as change from baseline on the ALS-FTD-Q. | endpoint or 24 months
  ALS-FTD-Q (Amyotrophic Lateral Sclerosis-Frontotemporal Dementia-Questionnaire) is a validated instrument for the screening of behavioral disturbances in ALS.
Clinical disease stage, defined as mean time spent in each stage of the King's and ALS Milano-Torino staging systems. | endpoint or 24 months
  The King's Staging Scale is a clinical staging system defining four stages of ALS assessed by way of a semi-structured interview with the participant.
Change from baseline in laboratory parameters: Urinary P75ECD (ectodomain of neurotrophin receptor p75), Neurofilament light and heavy chain, Plasma creatinine | endpoint or 24 months
  Plasma creatinine is assessed to monitor kidney function
Tolerability defined as time-to-discontinuation of assigned treatment since randomization | endpoint or 24 months
  the number of participants who discontinue study medication will be assessed to assess tolerability
Safety based on the safety assessments including neurological examinations, clinical laboratory evaluations, vital signs and frequency of adverse events (AEs) or serious adverse events (SAEs). | endpoint or 24 months
  (S)AEs will be categorized according to the Common Terminology Criteria for Adverse Events and will be rated for severity and association with study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Van den Berg, MD, Study Chair — TRICALS Foundation
Locations (13):
- Australia (6):
  - Flinders Medical Centre, Adelaide
  - Royal Brisbane and Women's Hospital, Brisbane
  - Calvary Health Care Bethlehem, Parkdale
  - Perron Institute, Perth
  - The University of Sydney (Royal prince Alfred hospital), Sydney
  - Concord hospital Sydney, Sydney
- University Hospital Leuven, Leuven, Belgium
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands
- Bellvitge University Hospital, Barcelona, Spain
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (3):
  - King's College Hospital, London
  - University College London Hospital NHS, London
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Undecided
Pending on privacy regulations.